CLINICAL TRIAL: NCT06062251
Title: Assessing the Performance of Shotgun Metagenomics in the Diagnosis of Complex Prosthetic Joint Infections (METAGENOS)
Brief Title: Assessing the Performance of Shotgun Metagenomics in the Diagnosis of Complex Prosthetic Joint Infections
Acronym: METAGENOS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC22.0208
Record Dates: First submitted 2023-09-25; First posted 2023-10-02 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Prosthetic Joint Infection
Keywords: Prosthetic joint infection; microbiological diagnosis; shotgun metagenomics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objectiveof this of a prospective, multicentre study is to evaluate the performance of shotgun metagenomics in the diagnosis of chronic Prosthetic joint infection (PJI) in comparison with the adapted MSIS diagnostic score..

The main questions it aims to answer are:

* To evaluate the performance of shotgun metagenomics in the diagnosis of chronic PJI in comparison with culture.
* To describe the epidemiology of bacterial species responsible for chronic PJI in Western France and their potential resistance to antibiotics.
* Analyzing the diagnostic performance of shotgun culture and metagenomics as a function of potentially administered antibiotic treatments A total of 143 patients sampled will be included. Six intraoperative samples will be taken for each patient, as part of routine care. In addition to the standard preoperative check-up, an extra volume of blood will be taken for CRP measurement at inclusion.

DETAILED DESCRIPTION:
Prosthetic joint infection (PJI) is one of the most serious and devastating complications of orthopaedic surgery, leading to a high risk of recurrence and disability, as well as increased mortality and management costs. Despite improvements in antibiotic prophylaxis procedures and surgical asepsis measures, the significant increase in the number of prostheses fitted worldwide has been accompanied by an increase in the number of infections. The infection rate has been estimated at between 1% and 2% after hip and knee arthroplasty.

Appropriate diagnosis and medical and surgical management of PJI are therefore essential to preserve and/or restore adequate motor function, minimise the risk of complications and prevent excessive morbidity. The microbiological diagnosis of PJI must be as early and exhaustive as possible in order to introduce rapid and effective antibiotic therapy and avoid the development of a biofilm (gangue around the material) or chronic infection (quiescent bacteria).

However, the diagnosis of PJI can be difficult to make in certain situations. Learned societies have established a definition of PJI and defined diagnostic scores combining clinical, biological, anatomopathological and cytological criteria. An initial definition was approved in 2011 by the Musculoskeletal Infection Society (MSIS). This definition was modified and subject to an international consensus review in 2013 (MSIS diagnostic score). In 2018, an international consensus meeting reviewed and adapted the MSIS score. This adapted score is more appropriate to current Medical Biology practices and to the non-accessibility of all diagnostic tests in laboratories (leucocyte esterase, alpha-defensin, ...).

In this definition of PJI, the positivity of 2 intra-operative samples to the same bacterial species is considered to be a major criterion. A wide range of bacteria can cause PJI: aerobic/anaerobic/intracellular/mycobacterial; somePJI can be polymicrobial. It is therefore essential to accurately identify these pathogens in order to administer appropriate antibiotic therapy and avoid chronicity of infection. Despite the optimisation of practices, culture of samples is negative in 5 to 30% of cases, despite the presence of diagnostic criteria for PJI. The most common causes are a lack of culture sensitivity, prior antibiotic administration and/or the presence of difficult or slow-growing pathogens. In these cases, intravenous broad-spectrum antibiotic therapy is administered, resulting in additional management costs, the occurrence of adverse treatment effects and the risk of acquiring resistance or intestinal dysbiosis.

In this context, "classic" molecular techniques are routinely used to overcome the limitations of culture for microbiological detection: bacterial-specific (including PCR targeting Staphylococcus aureus) or non-specific (bacterial universal PCR targeting the gene encoding 16S rDNA) (Figure 1). The latter approach was previously evaluated by the CRIOGO group (3Centre de Référence en Infections Ostéo-articulaires du Grand Ouest") with detection performance deemed disappointing in the context of PJI (sensitivity of 73.3%, specificity of 95.5%). Innovative molecular techniques for Next Generation Sequencing (NGS) are being developed, including shotgun metagenomics (sequencing of all the genetic material in a sample). Recent studies have evaluated the sensitivity of shotgun metagenomics in PJI, estimated at between 90.2% and 93.0% compared with bacterial culture and at around 95% compared with the MSIS diagnostic score.

However, these few recent studies evaluating shotgun metagenomics have only been carried out on a single sample per patient, which is insufficient according to the recommendations of the international and national consensuses on the management of PJI. In fact, four or even five intraoperative samples must be taken and analysed in microbiology to make the diagnosis of PJI. This high number of samples improves the sensitivity and completeness of bacterial detection and facilitates the interpretation of positive cultures for potentially contaminating skin bacteria (coagulase-negative Staphylococci, Cutibacterium acnes, etc.). To date, only one study has assessed the performance of shotgun metagenomics applied to several intraoperative samples per patient. Further studies are therefore needed to refine the performance of shotgun metagenomics in the context of PJI and to better assess the contribution of this costly technique, which requires considerable expertise to perform and interpret.

The setting up of a prospective, multicentre study in centres associated with the CRIOGO will make it possible to assess the performance of shotgun metagenomics in the management of chronic PJI. The performance of shotgun metagenomics will be assessed on the basis of four different samples per patient, in six centers specialising in the diagnosis of PJI, which makes the METAGENOS study unique compared with other studies. At the end of the project, the aim is to define the indications for using this innovative technique and to harmonise future regional practices.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years
* Patients being considered for surgery for suspected chronic PJI (time between joint replacement surgery and patient inclusion > 3 months)
* Social security affiliation
* No objection to participating in the study

Exclusion Criteria:

* Suspicion or documentation (positive blood cultures) of acute bacteremia at time of inclusion
* Patients under guardianship or trusteeship
* Pregnant or breastfeeding woman
* Patient deprived of liberty by legal or administrative decision
* Patients in psychiatric care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected chronic prosthetic joint infection
Sampling Method: Probability Sample
Enrollment: 143 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
PJI diagnosis | from samples taken during surgery. Shotgun metagenomics will be performed at the end of the inclusion of all patients, i.e. one year after the start of the study
  PJI diagnosis (positive/negative) obtained by shotgun metagenomics and by the adapted MSIS criteria (gold standard)MSIS diagnostic score (gold standard).

SECONDARY OUTCOMES:
PJI diagnosis (positive/negative) obtained by shotgun metagenomics and by culture | from samples taken during surgery. Shotgun metagenomics will be performed at the end of the inclusion of all patients, i.e. one year after the start of the study
Presence/absence of a bacterial species (by culture and/or shotgun metagenomics) in a patient sample considered infected according to the appropriate MSIS score | : from samples taken during surgery. Shotgun metagenomics will be performed at the end of the inclusion of all patients, i.e. one year after the start of the study
Resistance/sensitivity to antibiotics tested | immediate post-operative period (usually within 3-15 days following surgery)
PJI diagnosis (positive/negative) obtained by shotgun metagenomics and by culture in case of presence/absence of antibiotic therapy the month before surgery | from samples taken during surgery. Shotgun metagenomics will be performed at the end of the inclusion of all patients, i.e. one year after the start of the study

CONTACTS AND LOCATIONS:
Overall Officials: Rachel CHENOUARD, Dr, Principal Investigator — Angers HU; Stéphane CORVEC, PhD, Principal Investigator — Nantes HU; Chloé PLOUZEAU, Dr, Principal Investigator — Poitier HU; Sophie REISSIER, Dr, Principal Investigator — Rennes HU; Marie-Frédérique LARTIGUE, Dr, Principal Investigator — Tours HU
Locations (1):
- Brest university hospital, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: All collected data that underlie results in a publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.